CLINICAL TRIAL: NCT05869539
Title: A Phase I Trial of Adoptive Cell Therapy With Tumor-Infiltrating Lymphocytes and ANV419 in Patients With Advanced Melanoma. The BaseTIL-03M Trial
Brief Title: ACT-TIL and ANV419 for Advanced Melanoma.
Acronym: BaseTIL-03M
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Anaveon AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00575, th23laeubli
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Melanoma
Keywords: adoptive cell therapy; tumor-infiltrating lymphocytes; ANV419

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor-infiltrating lymphocyte transfer combined with ANV419 (Experimental): Patients have excisional biopsy/surgical resection of tumor lesion(s) (tumor collection) and TILs are expanded from this lesion/these lesions (TIL expansion).
  The transplant product will be produced in the Good Manufacturing Practice (GMP) facility of the University Hospital in Basel. TIL transfer to patient and first administration of ANV419 at day 0.
  Interventions: Drug: Combination of Tumor-infiltrating lymphocyte transfer with ANV419

INTERVENTIONS:
Drug: Combination of Tumor-infiltrating lymphocyte transfer with ANV419 — The study uses a personalized IMP (investigational medicinal product), i.e. TIL product in combination with ANV419.
  Day 0: Autologous TIL: (minimum 5 x 10^9 and up to 2x 10^11 lymphocytes) administered intravenously over 20 to 30 minutes.
  Day 0: Intravenous treatment with ANV419 at 243 μg/kg 2 hours after the TIL infusion. Actual body weight will be used to calculate the dose of ANV419.
  Day14: Intravenous treatment with ANV419 at 243 μg/kg. Actual body weight will be used to calculate the dose of ANV419.

SUMMARY:
In this study we aim to investigate safety and tolerability of tumor-infiltrating lymphocytes (TIL) adoptive cell therapy (ACT) incorporation in-vivo TIL expansion with ANV419 in patients with advanced melanoma

DETAILED DESCRIPTION:
In brief, this trial consists of four study periods: screening, pre-treatment, treatment, and observational follow-up.

In the screening period, patients are screened for trial eligibility. In the pre-treatment period, patients have excisional biopsy/surgical resection of tumor lesion(s) (tumor collection) and TILs are expanded from this lesion/these lesions (TIL expansion). Patients are permitted to receive bridging therapy outside of the study protocol.

In the treatment period, patients have TIL-ACT. TIL-ACT includes a detailed procedure of preparative chemotherapy, followed by transfer of the TIL product, followed by in-vivo TIL expansion with ANV419 (2 doses). TIL transfer is defined as day 0 in the study protocol. Patients have an End of Treatment visit (14 days after the last study treatment), a safety follow-up (30 days after the last study treatment) and an efficacy follow up, which is the End of Study visit (day +90).

Thereafter, patients will transfer to observational follow-up, which is conducted every 3 months until 1 year after TIL transfer.

Patients who terminate the study prematurely during any of the treatment period due to e.g., disease progression, toxicity, patient wish, etc. will also transfer to observational follow-up.

The regimen (TIL-ACT with ANV419) has not been tested. Review by the IDSMB (independent data safety monitoring board) will be performed after 3 patients (safety check).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following criteria will be eligible to participate in the study:

* Must provide written informed consent for the study.
* Must be able to comply with the study protocol as judged by the investigator.
* Are ≥ 18 years. 4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Have pathologically confirmed stage III (unresectable) or stage IV (metastatic) cutaneous melanoma, as per the American Joint Committee on Cancer staging system, 8th edition, and have experienced disease progression and exhausted all approved treatment option with curative intent.
* Have received at least one prior systemic treatment line of PD-(L)1 inhibitor and BRAF/MEK inhibition in case of BRAFV600 mutated melanoma. Adjuvant systemic treatment terminated ≥12 months prior to diagnosis of metastatic disease is not counted as a treatment line.
* Accessible tumor lesion(s) for TIL collection and willingness of the patient to undergo biopsy/resection of tumor lesion(s).
* Measurable disease as per RECIST v1.1 (following biopsy/resection of tumor lesion(s) for TIL collection).
* Adequate organ function (pulmonary, cardiovascular, hematological, hepatic, and renal function) per investigator's judgment. Cardiac stress testing is mandatory for all patients with underlying cardiac conditions and patients with age ≥50 years. 10. Female patients of childbearing potential must have a negative serum pregnancy test at the screening visit and a negative serum pregnancy test within 72 hours prior to start of preparative chemotherapy (day -7 in the study protocol).
* Female patients who are not postmenopausal, and who have not undergone surgical sterilization, must agree to use highly effective methods of contraception during the entire study period and for 6 months after the last dose of study drug. They must also agree not to donate eggs (ova, oocytes) during the same timeframe.
* Male patients with partners of childbearing potential must agree to use highly effective methods of contraception and barrier contraception (condom) during the entire study period and for 6 months after the last dose of study drug. They must also agree not to donate sperm during the same timeframe.

Exclusion Criteria:

* LDH (lactate dehydrogenase) ≥ 2x upper limit of normal (ULN).
* Life-expectancy ≤ 3 months per investigator's judgment.
* Have not recovered (i.e., ≤ Grade 1 or at baseline with the exception of alopecia or fatigue [up to Grade 2 allowed]) from immune-related adverse events (irAEs) resulting from prior immunotherapies. Patients who have endocrine immune-related AEs controlled by replacement therapy (i.e., hypothyroidism) due to previous treatment are eligible provided replacement therapy has been initiated and toxicity has returned to Grade 1.
* Have not recovered (i.e., ≤ Grade 1 or at baseline) from toxicities due to a previously administered chemotherapy, targeted small molecule therapy, or radiation therapy.

Note: If the patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study drug. Major surgery is defined as any surgery requiring entrance into a body cavity (e.g., chest, abdomen, or brain), organ removal, normal anatomy alteration, or joint replacement. Minor surgery is defined as any surgery in which skin, mucosa, or connective tissue sections are altered (e.g., biopsy, cataract, endoscopic procedures, etc.).

* Have been diagnosed with uveal/ocular or mucosal melanoma.
* Have a known additional malignancy (including all in-situ carcinoma) that is progressing or required active treatment within 2 years prior to enrollment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that have undergone potentially curative therapy and have no evidence of disease or in situ cervical cancer in patients who completed cancer-directed therapy or have evidence of stable disease and do not require active treatment.
* Have active central nervous system metastases and/or carcinomatous meningitis regardless of clinical stability. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to study treatment (day -7 in the study protocol), and any neurologic symptom has returned to baseline. New or enlarging brain metastases, as well as the use of steroids (≥10 mg of prednisone daily or equivalent) within the last 7 days prior to study drug are excluded.
* Have a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study treatment (day -7 in the study protocol).
* Are receiving systemic steroid ≥10 mg of prednisone daily or equivalent for any reason. Local steroid therapies (e.g., otic, ophthalmic, intra-articular, or inhaled medications) are acceptable. -
* Have an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. 11. Have a known history of, or any evidence of active, non-infectious pneumonitis.
* Have an active (measurable) and uncontrolled (unresponsive to current therapy) infectious disease (bacterial, fungal, viral, protozoic).
* Have a history of an acute coronary event (e.g., myocardial infarction) within 3 months prior to study treatment (day -7 in the study protocol), uncontrolled and symptomatic coronary artery disease, or congestive heart failure New York Heart Association Class III/IV.
* Have an average QTc interval > 470 msec at ECG-screening.
* Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or it is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 6 months after the last dose of study drug.
* Are known to be human immunodeficiency virus (HIV) positive (or tests positive for HIV 1 or 2 at Screening), unless the following criteria are met:

  1. Cluster of differentiation (CD)4+ lymphocyte count > 350 μL.
  2. Had no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the past 12 months.
  3. Have been on established anti-retroviral therapy for at least 4 weeks.
  4. Have an HIV viral load of > 400 copies/mL prior to study treatment (day -7 in the study protocol).

Note: Patients on strong cytochrome P450 (CYP)3A4 inhibitors or strong CYP3A4 inducers must be switched to an alternate effective anti-retroviral therapy regimen prior to study treatment or are excluded if regimen prior to study treatment cannot be altered.

* Have uncontrolled hepatitis B infection or hepatitis C infection. Note: Patients with hepatitis B (positive hepatitis B surface antigen) who have controlled infection (serum hepatitis B virus DNA by polymerase chain reaction that is below the limit of detection and receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of hepatitis B virus DNA. Note: Patients with hepatitis C (positive hepatitis C virus antibody) who have controlled infection (undetectable hepatitis C virus RNA by polymerase chain reaction either spontaneously or in response to a successful prior course of anti-hepatitis C virus therapy) are permitted.
* Have received a live vaccine within 30 days of study treatment (day -7 in the study protocol). Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Are positive for SARS-CoV2.
* Known hypersensitivity to any of the study therapies or drugs used for TIL production. - Any other conditions/diseases, dysfunctions, and/or findings, that would contraindicate the use of any of the study interventions or therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (%) | up to one year after TIL transfer
  Incidence of adverse events (%) will be recorded to assess safety of combination of Tumor-infiltrating lymphocytes with ANV419
Frequency of adverse events (number) | up to one year after TIL transfer
  Frequency of adverse events (number) will be recorded to assess safety of combination of Tumor-infiltrating lymphocytes with ANV419
Severity of adverse events (CTCAE v5.0 criteria) | up to one year after TIL transfer
  Severity of adverse events (CTCAE v5.0 criteria) will be recorded to assess safety of combination of Tumor-infiltrating lymphocytes with ANV419.
  CTCAE (Common Terminology Criteria for Adverse Events): Grade 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = fatal.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to one year after TIL transfer
  ORR is defined as the proportion of patients with a best overall response of partial response or better (assessed by the local investigators)
Duration of response (DOR) | up to one year after TIL transfer
  DOR is defined as the time from the first documented response and the date of the first documented tumor progression, death, or the last tumor assessment that occurred before subsequent therapy. DOR time for responders who have not progressed or died will be censored at the time of last tumor assessment
Progression-fee Survival (PFS) | up to one year after TIL transfer
  The progression-free survival (PFS) is defined as the time from registration to objective tumor progression (determined by local investigators), or death due to any cause, whichever occurred first. PFS time for patients who have not progressed or died will be censored at the time of the last tumor assessment
Overall survival (OS) | up to one year after TIL transfer
  OS is defined as the time from registration to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Läubli, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland